CLINICAL TRIAL: NCT02610569
Title: Comparison of the PillCamCOLON (C2) Capsule With Standard Endoscopy for the Evaluation of the Severity and the Endoscopic Healing of Patients With Ulcerative Colitis (UC)
Brief Title: Comparison of PillCamCOLON (C2) Capsule and Standard Endoscopy for the Evaluation of Patients With Ulcerative Colitis
Acronym: VCC2-RCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Arnaud Bourreille (Other)
Responsible Party: Sponsor-Investigator, Dr. Arnaud Bourreille, MD, Société Française d'Endoscopie Digestive
Organization: Société Française d'Endoscopie Digestive (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2013-A01674-41
Record Dates: First submitted 2015-04-27; First posted 2015-11-20 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis
Keywords: Colonic capsule; ulcerative colitis; mucosal healing; endoscopic score
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standart endoscopy (Active Comparator): Intervention: 2 standard endoscopy during anti-TNFalpha or vedolizumab treatment
  Interventions: Device: standard endoscopy
- PillCamCOLON (C2) (Experimental): Intervention : 2 PillCamCOLON (C2) during anti-TNFalpha or vedolizumab treatment
  Interventions: Device: PillCamCOLON (C2)

INTERVENTIONS:
Device: standard endoscopy — standard endoscopy will be either colonoscopy or rectosigmoidoscopy
  Arms: standart endoscopy
Device: PillCamCOLON (C2) — PillCamCOLON (C2) is a colon video-capsule
  Arms: PillCamCOLON (C2)

SUMMARY:
Ulcerative colitis (UC) is an inflammatory bowel disease progressing through flare-ups. The therapeutic objective, which was originally based on clinical remission, is currently evolving with the development of biotherapies towards the achievement of endoscopic remission. Current recommendations for therapeutic management advocate the achievement of endoscopic mucosal healing (EMH), with an observed decrease in the necessity for colectomy in the case of EMH. Endoscopic evaluation of the severity of UC is performed during a digestive endoscopy (colonoscopy for a complete colonic exploration, or recto-sigmoidoscopy for a partial exploration of the colon) from endoscopic activity scores adapted for UC.

Currently, the score the most commonly used is the MAYO endoscopic score. This is a global score of increasing intensity from 0 to 3, taking into account the following basic lesions: vascular pattern, granularity or/and friability of the mucosa, spontaneous bleeding, erosion and ulceration. However this score has limits: it does not distinguish deep cavitating ulcerations with mucous detachment from simple ulcerations which have a better prognosis.

A new endoscopic score specific for UC has been developed and is currently being validated. It is termed Ulcerative Colitis Endoscopic Index of Severity (UCEIS). This evaluation takes into account the three most reproducible factors - the vascular pattern, the presence of bleeding, and erosions or ulcerations including cavitating ulceration - in the total score.

To ensure optimal patient care and an adaptation of the therapeutic medical care to the endoscopic severity of the disease, endoscopic exploration should be performed recurrently. However, this exploration is an invasive procedure, requires general anaesthesia for colonoscopy, and can lead to potential complications such as perforation. This explains the poor acceptance by patients, resulting in a sub-optimal therapeutic support.

DETAILED DESCRIPTION:
For each patient, the study will be conducted in accordance with the following schedule:

Information/inclusion visit: D-30 (± 30 days)

* Full information about the trial
* Verification of inclusion and non-inclusion criteria
* Acquisition of informed consent (either the same day or after a period of reflexion)
* Medical and surgical history
* Clinical examination

Endoscopic visit: D0 On two consecutive days or within a maximum of seven days but obligatorily before the anti-Tumor Necrosis Factor (TNF) alpha treatment

* Faecal sample (calprotectin)
* Clinical examination
* Endoscopic examination by PillCamCOLON (C2) then by conventional endoscopy (colonoscopy)

  -The endoscopic examinations will each be analyzed by a different endoscopist working in a blinded evaluation. An UC activity score will be calculated depending on two scores: MAYO and UCEIS.
* Notification of Adverse Event (AE) / Serious Adverse Event (SAE)

Follow-up visit: W12 (12 weeks ± 5 days after D0)

* Faecal sample (calprotectin)
* Clinical examination
* Endoscopic examination by PillCamCOLON (C2) then by conventional endoscopy (coloscopy)

  -The endoscopic examinations will each be analyzed by a different endoscopist working in a blinded evaluation. An UC activity score will be evaluated depending on two scores: MAYO and UCEIS.
* Notification of AE/SAE

End-of-study visit (possibly by telephone) W14 (± 5 days)

*Notification of AE/SAE

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient between 18 and 70 years old
* Patient with UC requiring treatment with anti-TNFalpha or vedolizumab
* Patient affiliated to a social security scheme
* Patient able to understand and follow the study instructions
* Patient having signed an informed consent form

Exclusion Criteria:

* Patient with severe and acute colitis
* Patient with Crohn's disease or non-classified colitis
* Patient with an indication for surgical management of UC
* Patient with a history of sub-total or total colectomy, or with colostomy or ileostomy.
* Patient with a history of intestinal irradiation
* Patient with a known or suspected intestinal stricture
* Patient with clinical signs suggestive of intestinal stricture
* Patient with dysphagia with choking on solid food or swallowing disorders
* Patient with a contra-indication for an anti TNFalpha treatment
* Patient with a contra-indication for conventional endoscopy (colonoscopy or recto-sigmoidoscopy)
* Patient with congestive heart failure or severe renal impairment
* Patient with a pacemaker or other implanted electronic medical device
* Patient participating in another interventional clinical trial
* Pregnant or nursing woman
* Vulnerable individuals: persons deprived of liberty, under tutelage or guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Concordance between PillCamCOLON (C2) and conventional endoscopy for evaluation of the endoscopic MAYO score in patients with UC. | week 12 (W12)
  MAYO endoscopic score established by PillCamCOLON (C2) and conventional endoscopy of the common recto-colonic segment explored at week 12 (W12).

SECONDARY OUTCOMES:
Concordance between PillCamCOLON (C2) and conventional endoscopy for evaluation of the UCEIS score in patients with UC. | Week 12
  UCEIS endoscopic score established by PillCamCOLON (C2) and conventional endoscopy of the common recto-colonic segment explored at D0 and W12.
Concordance between PillCamCOLON (C2) and conventional endoscopy for measuring the variation of Mayo scores during an anti-TNF alpha or vedolizumab treatment | Week 12
  Mayo endoscopic scores established by PillCamCOLON (C2) and conventional endoscopy of the common recto-colic segment explored at D0 versus W12
Concordance between PillCamCOLON (C2) and conventional endoscopy for measuring the variation of the UCEIS scores during an anti-TNF alpha or vedolizumab treatment | Week 12
  UCEIS endoscopic scores established by PillCamCOLON (C2) and conventional endoscopy of the common recto-colic segment explored at W12
Presence of lesions upstream of the left colonic flexure using PillCamCOLON (C2), when recto-sigmoidoscopy is the conventional endoscopic procedure used. | Week 12
  Description of lesions located upstream of the left colonic flexure in terms of their localization and severity (in particular, ulcerations) visualized by PillCamCOLON (C2) when recto-sigmoidoscopy is the conventional endoscopic procedure used (at W12).
Capacity of PillCamCOLON (C2) to define endoscopic mucosal healing (MAYO score 0 and 1) as compared with recto-sigmoidoscopy, during treatment with anti-TNFalpha or vedolizumab. | Week 12
Correlation between calprotectin level in fecal sample and disease activity. | Week 12
  Calprotectin levels in fetal sample
Level of adequate colonic preparation during examinations with PillCamCOLON (C2). | Week 12
  Measurement of the quality of colonic preparation, relative to the commonly used scale, using all PillCamCOLON (C2) films obtained.
Reproducibility inter and intraobserver for the lesions' detection and for the severity grading by PillCamCOLON (C2) | Week 12
  Reproducibility inter and intraobserver concerning the lesions descriptions and their severity.
Analog visual scale (AVS) the preference of the patients and their acceptability of each of 2 examinations | Week 12
  AVS on exams acceptability between PillCamCOLON (C2) and conventional endoscopy
Adverse events due to PillCamCOLON (C2) and conventional endoscopy | Week 14
  To evaluate the tolerance of these two endoscopic examination procedures. Adverse events due to PillCamCOLON (C2) and adverse events due to conventional endoscopy.
Capacity of PillCamCOLON (C2) to define the extent of UC, as compared with colonoscopy | Week 12
Percentage of complete exploration by PillCamCOLON (C2) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourreille, MD, Principal Investigator — University Hospital of Nantes
Locations (1):
- University Hospital of Nantes, Nantes, France